CLINICAL TRIAL: NCT06359418
Title: Acupuncture for Prediabetes With Combined Obesity: a Multicenter Randomized Controlled Trial
Brief Title: Acupuncture for Prediabetes With Combined Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Guangdong Provincial Hospital of Chinese Medicine, Zhuhai (Unknown); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Linyi Hospital of Traditional Chinese Medicine (Unknown); The Second Affiliated Hospital of Guizhou University of Traditional Chinese Medicine (Unknown); Xi'an Traditional Chinese Medicine Hospital (Other); Qingdao Traditional Chinese Medicine Hospital (Unknown); Xi'an Hospital of Traditional Chinese Medicine (Other); Heilongjiang Academy of traditional Chinese Medicine (Unknown); The Affiliated Hospital of Qingdao University (Other); Yantai Hospital of Traditional Chinese Medicine (Unknown); Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-007-KY
Record Dates: First submitted 2024-03-24; First posted 2024-04-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Abdominal Obesity; PreDiabetes
Keywords: acupuncture; randomized controlled trial; Obesity; Abdominal Obesity; PreDiabetes
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Prediabetic State | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The participants in the acupuncture group will receive treatment that consists of 28 acupuncture sessions over a 12-week (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 8 weeks) period after baseline, each for 30 minutes. Hwato brand disposable acupuncture needles (size 0.30 x75mm; size 0.30 x 50mm; size 0.30 x 40mm) will be used. BaiHui(DU20), YinTang(EX-HN3), ShuaiGu(GB8), QuChi ( LI11), ZhongWan(RN12), XiaWan(RN10), TianShu(ST25), GuanYuan(RN4), FengLong(ST40), Daimai(GB26) and Fujie(SP14) were selected as acupoints protocol.
  At the same time, all participants will receive standardized lifestyle intervention counseling from randomization to end of whole study period, about once a month. Participants were advised to achieve a reduced-calorie diet (500-kcal deficit per day relative to the energy expenditure estimated at the time they underwent randomization) and increased physical activity (with 150 minutes per week of physical activity).
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): The participants in the sham acupuncture group will receive shallow needling at sham DU20, EX-HN3, GB8, LI11, RN12, RN10, ST25, RN4, ST40, GB26 and SP14. The protocol includes the same duration and frequency of sessions as for the acupuncture treatment, but the treatment was delivered superficially at non-acupuncture points 10-20 mm to the lateral of corresponding acupuncture and not above a meridian line. The Hwato brand disposable acupuncture needles(size 0.20 x25mm) will be inserted.
  At the same time, all participants will receive standardized lifestyle intervention counseling from randomization to end of whole study period, about once a month. Participants were advised to achieve a reduced-calorie diet (500-kcal deficit per day relative to the energy expenditure estimated at the time they underwent randomization) and increased physical activity (with 150 minutes per week of physical activity).
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — The acupuncture needle (size 0.30x40mm) will be inserted into DU20, EX-HN3 and GB8 acupoints at the depth of 15-30mm; The acupuncture needle (size 0.30x50mm or size 0.30x75mm) will be inserted into other acupoints at the depth of 40-70mm; Manipulation will be done after insertion (6 times of small amplitude and uniform twist).
  Arms: Acupuncture
Device: Sham acupuncture — The acupuncture needle (size 0.20x25mm) will be inserted into all acupoints at the depth of 2mm without any manipulation.
  Arms: Sham acupuncture

SUMMARY:
The clinical trial aims to evaluate the efficacy and safety of acupuncture in reducing weight and waist circumference while modulating glucose and lipid metabolism in Prediabetes with Combined Obesity.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects are eligible to be included in the trial only if all of the following criteria apply:

1. Simultaneously meeting the diagnostic criteria for both general obesity, abdominal obesity, and prediabetes;
2. Aged 18-64 years old;
3. Informed consent obtained before any trial-related activities.

Exclusion Criteria:

-

Subjects are excluded from the trial if any of the following criteria apply:

1. Obesity of known endocrine origin (e.g., untreated hypothyroidism, Cushing's syndrome, established Polycystic Ovary Syndrome);
2. impaired glucose regulation due to hyperthyroidism, endocrine tumors and extensive liver damage;
3. Diagnosis of type 1 or type 2 diabetes per the judgment of the investigator;
4. Current or history of treatment with medications that may cause significant weight gain, within 3 months prior to screening, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), antidepressants, antipsychotic, mood stabilizers, antiepileptic and hormone contraceptive;
5. History of pancreatitis or pancreatectomy;
6. Previous or planned (during the trial period) obesity treatment with surgery or a weight-loss device;
7. Current participation (or within the last month) in an organized weight reduction program or currently using or used medication for obesity or hyperglycemia within 3 months before screening: liraglutide, exenatide, pramlintide, orlistat, topiramate, phenteremine, or metformin (either by prescription or as part of a clinical trial);
8. A self-reported change in body weight >5 kg within 3 months before screening irrespective of medical records;
9. Serious medical conditions (including but not limited to ongoing renal or hepatic insufficiency, congestive heart failure, myocardial infarction, stroke, hematopoietic system diseases, progressive malignant tumor or other serious consumptive diseases); history of angina pectoris, transient ischemic attack, claudication, or acute limb ischemia within the past 6 months prior to screening;
10. Serious psychiatric illness, including lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, and anorexia nervosa; current serious personality disorder, (e.g. borderline or antisocial), current severe major depressive disorder, recent (previous 6 months) suicide attempt or current active suicidal ideation, recent hospitalization due to psychiatric illness;
11. Skin infection, blood coagulation disorders and other conditions that are not suitable for acupuncture;
12. Metal allergies or severe fear of needles;
13. Pregnant or breast-feeding women or planning to become pregnant during the study period;
14. Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
The percentage change in body weight from baseline to week 12 | week 12
  The weight is measured by electronic scale with an accuracy of 0.1kg.
The percentage change in waist circumference from baseline to week 12 | week 12
  The waist circumference is measured by a fiberglass tape measure with an accuracy of 0.1 centimeters.

SECONDARY OUTCOMES:
The percentage change in body weight compared to the baseline | week 4, week 8, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  The weight is measured by electronic scale with an accuracy of 0.1kg.
The percentage change in waist circumference compared to the baseline | week 4, week 8, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  Waist circumference measurements are accurate to 0.1cm.
Achievement of a reduction in body weight of 5% or more compared to the baseline | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  A 5% reduction is the weight loss target for obese patients recommended in most guidelines.
Achievement of a reduction in body weight of 7% or more compared to the baseline | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  A 7% reduction is a weight loss target for obese patients with other metabolic diseases recommended in most guidelines.
The change in body weight from baseline | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  The weight is measured by electronic scale with an accuracy of 0.1kg.
The change in waist circumference from baseline | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  Waist circumference measurements are accurate to 0.1cm.
The proportion of participants reverting to normoglycaemia | week 12, week 36, week 52
  The determination is based on the results of blood glucose laboratory parameters.
The proportion of participants developing diabetes | week 12, week 36, week 52
  The determination is based on the results of blood glucose laboratory parameters.
The change in 2hPG from baseline and percentage of patients who returned to normal | week 12, week 36, week 52
  2hPG, 2-hour post-load Plasma Glucose, will be measured by oral glucose tolerance test, in mmol/L.
The change in FPG from baseline and percentage of patients who returned to normal | week 12, week 36, week 52
  FPG is fasting plasma glucose, the result will be reported in mmol/L.
The change in HbA1c from baseline and percentage of patients who returned to normal | week 12, week 36, week 52
  HbA1c is glycated haemoglobin, the result will be reported in percentage (%) units.
The change in 1hPG from baseline and percentage of patients who returned to normal | week 12, week 36, week 52
  1hPG, 1-hour post-load Plasma Glucose, will be measured by oral glucose tolerance test, in mmol/L.
Changes in appetite VAS score from baseline | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  VAS=visual analogue scale; The VAS of appetite is a 100mm with two ends pointing to "none" and "difficult to control", respectively, and the subjects mark them on the online segment according to their perception. Appetite is quantitatively evaluated by measuring the distance from the left side of the segment to the marked point.
The change in BMI from baseline | week 4, week 8, week 12, week 16, week 24, week 36, week 52
  BMI=Body Mass Index, weight and height will be combined to report BMI in kg/m^2.
The change in WHR from baseline | week 4, week 8, week 12, week 16, week 24, week 36, week 52
  WHR=Waist-to-Hip Ratio, the ratio of waist to hip circumference, waist and hip circumference are accurate to 0.1cm.
The change in WHtR from baseline | week 4, week 8, week 12, week 16, week 24, week 36, week 52
  WHtR=waist-to-Height Ratio, the ratio of waist circumference to height. Both are in cm units, accurate to 0.1cm.
The change in FINS from baseline | week 12, week 36, week 52
  FINS is fasting insulin, the result will be reported in pmol/L.
The change in HOMA-IR from baseline | week 12, week 36, week 52
  HOMA, Homeostatic Model Assessment, is a mathematical model reflecting the interaction of glucose and insulin in different organs (including pancreas, liver, and surrounding tissues). lt was first proposed by Matthews in 1985. Insulin Resistance (HOMA-IR) will be evaluated by fasting plasma glucose (FPG) and fasting insulin (FlNS). The calculation method is HOMA-IR=FPG xFINS/22.5.
The change in HOMA-β from baseline | week 12, week 36, week 52
  HOMA, Homeostatic Model Assessment, is a mathematical model reflecting the interaction of glucose and insulin in different organs (including pancreas, liver, and surrounding tissues). lt was first proposed by Matthews in 1985. Islet β cell function (HOMA-β ) will be evaluated by fasting plasma glucose (FPG) and fasting insulin (FlNS). The calculation method is HOMA- β = 20 x FINS/ (FPG-3.5).
The change in Serum total cholesterol from baseline | week 12, week 36, week 52
  The Serum total cholesterol will be reported in mmol/L.
The change in Triglyceride from baseline | week 12, week 36, week 52
  The Triglyceride will be reported in mmol/L.
The change in Low-Density Lipoprotein Cholesterol from baseline | week 12, week 36, week 52
  The Low-Density Lipoprotein Cholesterol will be reported in mmol/L.
The change in High-Density Lipoprotein Cholesterol from baseline | week 12, week 36, week 52
  The High-Density Lipoprotein Cholesterol will be reported in mmol/L.
The change in Serum Uric Acid from baseline | week 12, week 36, week 52
  The Serum Uric Acid will be reported in μmol/L.
The change in C-reactive protein from baseline | week 12, week 36, week 52
  The C-reactive protein will be reported in mg/L.
The change in blood pressure from baseline | week 4, week 8, week 12, week 16, week 24, week 36, week 52
  Record the values of systolic blood pressure and diastolic blood pressure in mmHg.
Changes of the score of the European five-dimensional Health scale (EQ-5D-5L) compared with the baseline. | week 12, week 36
  EQ-5D-5L=European Quality of Life Five Dimension Five Level Scale Questionnaire. The questionnaire which is widely used to evaluate the quality of life of the general population is divided into two parts: EQ-5D health description system and EQ-VAS. The score was calculated by calculating formula according to the choices made by the subjects in the questionnaire.
Changes of the PHQ-4 score from the baseline. | week 12, week 36
  PHQ-4=patient health questionnaire-4. PHQ-4 consists of the first two items in PHQ-9 (PHQ-2) and the first two items in GAD-7 (GAD-2), including depression and anxiety. It is translated into Chinese by scholars and verified by scholars. It has good reliability and validity and is suitable for depression and anxiety screening.

OTHER OUTCOMES:
Expectance assessment | baseline
  Participants will be asked the following question: What do you think will happen to your obesity and prediabetes in 3 months?
Assessment of belief in acupuncture | baseline
  Participants will be asked to answer "do you think acupuncture is helpful for obesity and prediabetes?" And three other related questions.
Blinding assessment | week 12
  Participants will be asked the following question: do you think you have received traditional acupuncture in the past weeks?
Safety assessment | week 0 to week 52
  Adverse events and severe adverse events will be recorded in the case report form, whether related to interventions ol not.
Adherence assessment of acupuncture | weeks 1 to week 12
  Adherence will be assessed via counting treatment sessions. Those who complete over 80% treatment sessions will be defined as of good adherence.
Adherence assessment of life modification | week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 52
  Adherence will be assessed through dietary diaries and physical activity questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China